CLINICAL TRIAL: NCT05760430
Title: A Single-center Study of the Synergistic Effect of Portal Venous Supply Control and Immunotherapy in Hepatocellular Carcinoma
Brief Title: The Synergistic Effect of Portal Venous Supply Control and Immunotherapy in Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-0857
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2022-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Portal Venous Supply Control; Immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): After cTACE, 3 mg/kg of Camrelizumab was injected intravenously once every three weeks+250 mg of Apatinib mesylate tablets were taken orally once a day. PVE was performed on the half liver with the largest tumor load 2 weeks after CTACE.
  Interventions: Combination Product: PVE+cTACE+Camrelizumab+Apatinib
- Control group (Active Comparator): After cTACE, 1200 mg of Atirizumab+15 mg/kg of Bevacizumab was injected intravenously every three weeks.
  Interventions: Combination Product: cTACE+Atirizumab+Bevacizumab

INTERVENTIONS:
Combination Product: PVE+cTACE+Camrelizumab+Apatinib — After cTACE, 3 mg/kg of Camrelizumab was injected intravenously once every three weeks+250 mg of Apatinib mesylate tablets were taken orally once a day. PVE was performed on the half liver with the largest tumor load 2 weeks after CTACE.
  Arms: Experimental Group
Combination Product: cTACE+Atirizumab+Bevacizumab — After cTACE, 1200 mg of Atirizumab+15 mg/kg of Bevacizumab was injected intravenously every three weeks.
  Arms: Control group

SUMMARY:
Hepatocellular carcinoma is one of the most common solid malignant tumors. The prognosis of unresectable hepatocellular carcinoma is very poor. According to the current literature and the clinical practice of our center, portal vein blood supply control may have great potential in the synergistic treatment of unresectable hepatocellular carcinoma. Thus, we hope to study the safety and efficacy of portal blood supply control +TACE+ Camrelizumab + Apatinib combined therapy in initial unresectable hepatocellular carcinoma through a single-center clinical trial, and explore the synergistic effect of portal blood flow control in target immune therapy of hepatocellular carcinoma.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the most common solid malignant tumors and the main cause of cancer-related deaths worldwide. The main treatment method for patients with unresectable or advanced HCC (such as patients with vascular invasion, distant metastasis, or tumor-related symptoms) is systemic therapy such as immunotherapy combined with targeted drugs. The median OS of patients treated with first-line bevacizumab (T)+atilizumab (A) was 19.2 months, and the ORR was 30%; The median OS was 22 months and the ORR was 36% when the Lenvatinib+Pembrolizumab (K-drug) regimen was used in the second-line treatment of patients with unresectable HCC. At present, the combination of domestic PD-L1 monoclonal antibody, Camrelizumab, and VEGFR-2 inhibitor, Apatinib, shows great potential in the treatment of Chinese patients with unresectable HCC. Phase II data shows that the ORR, DCR, mPFS, and mOS for first-line treatment are 34%, 77%, 5.7 months, and 20.3 months respectively.

However, the benefits for patients are still very limited, and the clinical treatment of non-resectable HCC is facing serious challenges. Therefore, it is necessary to take a reasonable multidisciplinary comprehensive treatment strategy, to establish a new effective treatment plan and further improve the prognosis and quality of life of patients.

The anti-vascular treatment of HCC is the basis of immunotherapy and an important trigger and intensifier. The reason and mechanism are that hepatocellular carcinoma can be secondary to liver injury caused by various reasons, such as chronic alcohol consumption, chronic hepatitis B and C infection, non-alcoholic fatty liver, etc., but all of them are manifested by increased blood vessels and significant vascular abnormalities, which suggests that blood supply plays an important role in the occurrence and development of HCC. A large number of targeted anti-vascular drugs have been used in the treatment of hepatocellular carcinoma. Angiogenesis inhibitors can specifically inhibit VEGF-mediated dendritic cell maturation disorder, promote antigen presentation and T cell immune response to tumor antigen; At the same time, it antagonizes angiogenesis, blocks tumor blood supply, normalizes tumor blood vessels, and increases T cell infiltration in tumor cells.

The hepatic artery is the main blood supply source of the tumor, so angiogenesis inhibitors often combine with TACE to directly and effectively block the blood supply of the tumor, which can not only effectively inhibit angiogenesis around the tumor, but also delay the progress of tumor and thus improve the effect of tumor treatment. It is noteworthy that portal vein blood flow also plays an important role in the occurrence and development of HCC.

Angiogenesis inhibitors can directly or indirectly affect the portal vein blood flow and improve the prognosis. It has been reported in the literature that angiogenic inhibitors such as sorafenib and lenvatinib can significantly reduce portal vein pressure and effectively prolong the survival period of advanced HCC.

Multiple blood supply blockages also show certain therapeutic significance. In post-line treatment, dual/multiple anti-vascular therapies show therapeutic effects. For example, the multi-target anti-vascular drug regorafenib can be used as the second-line drug after the first-line treatment of sorafenib. The median survival period of sorafenib+regorafenib second-line treatment is 24 months.

The response rate of targeted immunotherapy is higher in advanced patients with portal vein tumor thrombus. Not only does the tumor focus shrink, but the tumor thrombus also shrinks or even disappears. This may be because the lack of blood supply in the portal vein further reduces the blood supply of the tumor and tumor thrombus, thus promoting the response to systemic therapy.

In our previous clinical practice and research, we found that the control of portal vein blood flow on the affected side may have synergistic anti-tumor effects. The advanced patients treated with targeted immunotherapy combined with portal vein blood supply control, such as portal vein embolization (PVE), showed a good treatment response. In the future, while the volume of the residual liver increased, the tumor focus was significantly reduced. The patients obtained the opportunity of surgical resection, and some patients even achieved complete response (CR).

Embolization of the portal vein of the affected liver segment leads to an increase in the blood supply of the residual liver in the future, and realizes a rapid increase in the volume of the residual liver in the future, so as to ensure the quality and prognosis of hepatectomy, which is a common method for patients with early liver cancer before hepatectomy.

At present, there is no study on the use of a portal vein blood supply control combined system for the treatment of unresectable HCC conversion. Based on the current research and clinical practice, we propose a hypothesis that strengthening blood supply control is conducive to the conversion treatment of HCC, and controlling the blood supply of the portal vein has an important synergistic effect on the treatment of unresectable HCC. Portal vein blood supply control combined with TACE and targeted immunotherapy can further enhance the conversion rate of unresectable HCC, bring more opportunities for patients' subsequent surgery or local treatment, and help to prolong the survival period of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female aged ≥ 18;
2. Primary hepatocellular carcinoma confirmed by pathology;
3. There is no extrahepatic metastasis and portal vein tumor thrombus (Barcelona stage b), which cannot be removed after the evaluation of the surgeon, but there is a potential surgical opportunity after the tumor is significantly reduced;
4. Have not received treatment in the past;
5. At least 1 measurable lesion meeting the RECIST v1.1 or mRECIST standard;
6. Liver function is Child-Pugh A;
7. ECOG PS 0~1 before entering the group;
8. Organs and bone marrow are fully functional:

9 Expected survival period ≥ 3 months; 10. Women of childbearing age who have not undergone surgical sterilization should take effective contraceptive measures within 3 months from enrollment to the end of the trial; 11. Sign a written informed consent and be able to comply with the visit and relevant procedures specified in the plan.

Exclusion Criteria:

1. The patient has any history of active autoimmune disease or autoimmune disease;
2. The patient is using immunosuppressant or systemic hormone therapy to suppress immune function;
3. Known central nervous system metastasis or hepatic encephalopathy;
4. Severe allergic reaction to other monoclonal antibodies;
5. Have a history of organ transplantation;
6. The patient has the serious basic disease and cannot tolerate treatment;
7. The patient has previously received other anti-PD-1 antibody treatment or other anti-PD-1/PD-L1 immunotherapy, or has previously received apatinib treatment;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Conversion rate | The time frame is from the first treatment to the last treatment, an average of 2 years.
  The proportion of patients with unresectable hepatocellular carcinoma who have achieved surgical R0 resection after combined treatment.

SECONDARY OUTCOMES:
Objective response rate | The time frame is from the first treatment to the last treatment, an average of 2 years.
  The proportion of hepatocellular carcinoma patients with complete and partial remission in all evaluable patients.
Residual liver volume proliferation rate after hepatectomy | The time frame is from the first treatment to the last treatment, an average of 2 years.
  The proportion of residual liver volume to the preoperative liver volume of the patient was measured by CT image.
Progression-free survival | The time frame is from the first treatment to the last treatment, an average of 2 years.
  The time from the first treatment to the first assessment of recurrence, metastasis or death.
Time to progress | The time frame is from the first treatment to the last treatment, an average of 2 years.
  The time from the first treatment to the first assessment of recurrence or metastasis.
Overall survival | The time from the first treatment to death (up to 3 years). The last follow-up time is for the patients who lost the follow-up, and the end of the follow-up is for the patients who are still alive at the end of the study.
  The time from the first treatment to death (up to 3 years). The last follow-up time is for the patients who lost the follow-up, and the end of the follow-up is for the patients who are still alive at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Yan, Dctor, Study Chair — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available from the author on reasonable request.